CLINICAL TRIAL: NCT00555776
Title: Phase 2 Effect of Gabapentin on Idiopathic Subjective Tinnitus
Brief Title: Effect of Gabapentin on Idiopathic Subjective Tinnitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Islamic Azad University of Mashhad (Other)
Responsible Party: Dr.Mahboobeh Adami Dehkordi, Assisstant professor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gaba-tinntus-145
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2009-01-06 (Estimated); Status verified 2008-08

CONDITIONS: Subjective Tinnitus
Keywords: tinnitus; gabapentin
MeSH Terms: conditions — Tinnitus | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Randomly,half of the subjects are given Gabapentin.
  Interventions: Drug: Gabapentin
- 2 (Placebo Comparator): Randomly,half of the subjects receive placebo.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Gabapentin — Gabapentin, 600 mg bid for the first two weeks, increased to a maximum dose of 1800 mg per day during the next 6 weeks if necessary.
  Other Names: Neurontine
  Arms: 1
Drug: placebo — placebo is given with the same definition as Gabapentin
  Arms: 2

SUMMARY:
The purpose of this study is to determine wether Gabapentin which is useful for treating neuropathic pains, is effective on idiopathic subjective tinnitus.

DETAILED DESCRIPTION:
Tinnitus is the perception of sound in the absence of acoustic stimulation. It can be subjective or objective. .

Despite numerous researches,no effective treatment for people who suffer from tinnitus has yet been stablished.

As there are many evidences suggesting that loss of inhibition in the central nervous system may be responsible for many aspects of auditory dysfunction,including tinnitus; and as Gabapentin (Neurontin), a gama-aminobutyric acid (GABA) analogue, is an effective medication in conditions where inhibition in the CNS is impaired; we guess that Gabapentin might be useful for treating idiopathic subjective tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* patients with subjective idiopathic tinnitus

Exclusion Criteria:

* tinnitus with known underlying cause
* pregnant women and patients younger than 18 or older than 75 years
* patients with impaired renal function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-04 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Reduction in the sensation of Tinnitus by the patient or complete resolution of tinnitus;by the patient's scoring it from one to ten, before and after prescribing Gabapentin. | two months

SECONDARY OUTCOMES:
Relieve of complications of tinnitus, such as sleep difficulties. | two months

CONTACTS AND LOCATIONS:
Overall Officials: Mahboobeh Adami Dehkordi, MD, Principal Investigator — ENT department of Mashhad azad university of mashhad
Locations (1):
- ENT department of Mashhad Azad medical university, Mashhad, Khorasan Razavi, Iran

REFERENCES:
- [Result] Bakhshaee M, Ghasemi M, Azarpazhooh M, Khadivi E, Rezaei S, Shakeri M, Tale M. Gabapentin effectiveness on the sensation of subjective idiopathic tinnitus: a pilot study. Eur Arch Otorhinolaryngol. 2008 May;265(5):525-30. doi: 10.1007/s00405-007-0504-9. Epub 2007 Oct 25. PMID 17960408